CLINICAL TRIAL: NCT07255495
Title: Effects of Neuromuscular Scoliosis Surgery on Nutritional Metabolism
Acronym: SORONOUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL25_0018
Record Dates: First submitted 2025-08-25; First posted 2025-12-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy; Scoliosis
Keywords: energy metabolism; quality of life; nutritional support
MeSH Terms: conditions — Cerebral Palsy; Scoliosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of group before and after spinal surgery (Experimental): Assessment of food intake, body composition, energy expenditure, quality of life, achievement of customized goals before and after spinal surgery
  Interventions: Diagnostic Test: Absorptiometry and indirect calorimetry; Behavioral: Questionnaires

INTERVENTIONS:
Diagnostic Test: Absorptiometry and indirect calorimetry — Assessment of body composition with dual-energy absorptiometry : 1 month before surgery and 6 months after surgery
  Assessment of energy expenditure with indirect calorimetry : 1 month before surgery and 6 months after surgery
Behavioral: Questionnaires — Assessment of food intake with a standardized questionnaire : 6 months before surgery, 1 month before surgery, 3 months after surgery and 6 months after surgery
  Assessment of quality of life with the CP Child Score questionnaire : 6 months before surgery, 1 month before surgery, 3 months after surgery and 6 months after surgery
  Assessment of the achievement of customized goals established one month before the scoliosis surgery : 3 months after surgery and 6 months after surgery

SUMMARY:
Cerebral palsy is the primary cause of disability in France. It is a non-progressive condition leading to movement and posture troubles, but also to cognitive and sensory problems. Spasticity is one of the most regular consequences. It leads to a muscular failure with permanent contractions. Muscular dysfunction can generate scoliosis (in 60% of cases). Scoliosis can lead to pain, sitting difficulties (with chances of bedsores), and cardiopulmonary complications.

These children often have cachexia (eating difficulties, trouble with deglutition). It leads to a weakening of their immune defenses, which favors post-operative infections, a weakening of their respiratory muscles, and circulatory difficulties with negative effects on scarring. Cachexia is a pessimistic prognosis.

A back brace can be used to contain the scoliosis but never cures it. Another option for treating this affection would be surgery. Surgery is another treatment. It consists in straightening and holding the spine with metal rods, held by vertebral anchors placed at both ends of the scoliosis. Surgery is the gold standard.

Surgery induces risks such as bleeding, healing complications and infection. The probability to face complications increases with malnutrition.

The first hypothesis is that surgery could improve the nutrients intakes and the weight of the patient.

The investigators also believe that it could improve the patient's body composition (body fat and lean mass) and their basic metabolic rate.

The third hypothesis is that surgery-involved changes (nutrition enhancement, sitting improvement, decrease of respiratory work) could lead to an improvement of the patient's quality and life and respiratory functions.

The SORONOUS project aim to prove the benefits of this surgery from a nutritional and from a general point of view in order to help make the surgical decision and avoid any care delay. In addition, it aim to identify and quantify the post-operative weight gain; while providing us with a better understanding of the behavior of pre-operative cachexia among these patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cerebral palsy
* Subjects between 10 and 20 years old
* Neuromuscular scoliosis requiring surgical care (accepted by the patient or their legal representatives)
* Subjects escaping scoliosis treatment with a brace

Exclusion Criteria:

* History of spine surgery
* Impossible follow-up during the study time
* Peripheral or non spastic palsy
* Palsy caused by a medullary injury
* Subject with a contraindication to DXA scan examination (e.g. coronary stents or cardiac metal sutures, pacemaker or automatic defibrillator)
* Absence of voluntary and informed consent signed by the patient or their legal representatives
* Patient or their legal representatives with no social security affiliation
* Patient or their legal representatives deprived of freedom by a judicial or administrative decision
* Pregnant, laboring, or breastfeeding woman

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Dietary intakes modifications before and after scoliosis surgery | Between 1 month before surgery and 6 months after surgery
  Assessment of the dietary intakes in kcal/day (dietary intakes per os and/or gastrostomy and/or nasogastric tube) by nutrition questionnaires and based on the average food intake over the last 7 days. Caregivers will provide information on food intake for each day and each meal during the seven days preceding the consultation using a food intake sheet. A standardized table will be used to calculate the equivalents between food intake and energy intake (kcal). An average will be calculated over the 7 days to obtain a dietary intake in kcal/day. Comparison of the dietary intakes between one month before scoliosis surgery and six months after surgery

SECONDARY OUTCOMES:
Dietary intakes modifications before and after scoliosis surgery | Between 1 month before surgery and 3 months after surgery
  Assessment of the dietary intakes in kcal/day (dietary intakes per os and/or gastrostomy and/or nasogastric tube) by nutrition questionnaires and based on the average food intake over the last 7 days. Caregivers will provide information on food intake for each day and each meal during the seven days preceding the consultation using a food intake sheet. A standardized table will be used to calculate the equivalents between food intake and energy intake (kcal). An average will be calculated over the 7 days to obtain a dietary intake in kcal/day. Comparison of the dietary intakes between one month before scoliosis surgery and six months after surgery
Weight comparison before and after scoliosis surgery | Between 1 month before surgery and 6 months after surgery
  Weight measurement in kilograms of each participant. Weight comparison between one month before surgery and six months after surgery
Weight comparison before and after scoliosis surgery | Between 1 month before surgery and 3 months after surgery
  Weight measurement in kilograms of each participant. Weight comparison between one month before surgery and three months after surgery
Assessment of the quality of life before and after scoliosis surgery | Between 1 month before surgery and 6 months after surgery
  Assessment of the quality of life, comfort, transfers and mobility with the CP Child Score questionnaire (Caregivers' Priorities and Child Health Index of Life with Disabilities). Each domain and the total score are standardized on a scale from 0 to 100. Higher scores indicate better comfort, function, and well-being of the child as perceived by the caregiver.
  Comparison of the 1 month before surgery and 6 months after surgery scores
Assessment of the quality of life before and after scoliosis surgery | Between 1 month before surgery and 3 months after surgery
  Assessment of the quality of life, comfort, transfers ad mobility with the CP Child Score questionnaire (Caregivers' Priorities and Child Health Index of Life with Disabilities). Each domain and the total score are standardized on a scale from 0 to 100. Higher scores indicate better comfort, function, and well-being of the child as perceived by the caregiver.
  Comparison of the 1 month before surgery and 3 months after surgery scores
Change of respiratory rate before and after surgery | Between 1 month before surgery and 6 months after surgery
  Assessment of the respiratory rate (breaths per minute) through clinical examination.
  Comparison of the respiratory rate between one month before surgery and six months after surgery
Change of respiratory rate before and after surgery | Between one month before surgery and three months after surgery
  Assessment of the respiratory rate (breaths per minute) through clinical examination.
  Comparison of the respiratory rate between one month before surgery and six months after surgery
Change of metabolic rate before and after surgery | Between 1 month before surgery and 6 months after surgery
  Quantification of the basic metabolic rate (kcal/d) with indirect calorimetry (inhalation chamber or gas mask). Comparison of the metabolic rate one month before surgery and six months after surgery
Change of weight distribution before and after surgery | Between one month before surgery and six months after surgery
  Assessment of the body composition with dual-energy absorptiometry (DEXA scan). The body composition, including body fat (kg, %) and lean mass (kg, %) will be assessed on the whole body and on different body segments (upper limbs, lower limbs and trunk).
  Comparison of the body composition one month before surgery and six months after surgery
Assessment of the achievement of customized goals established one month before the scoliosis surgery | 3 months after surgery
  Specific customized goals will be established one month before surgery with the Goal Attainment Scale. The goals will concern several aspects of daily life (e.g. to dress up, to brush your teeth). The initial Goal is set at -2 point scale. on Each goal is rated on a 5-point scale: Much less than expected (-2); Somewhat less than expected (-1) ; Expected level of achievement (0); Much more than expected outcome (+2), Somewhat more than expected (+1). A higher score (closer to +2) indicates a better outcome, meaning the goal was achieved beyond expectations. Assessment of the achievement of these goals three months after surgery
Assessment of the achievement of customized goals established one month before the scoliosis surgery | 6 months after surgery
  Specific customized goals will be established one month before surgery with the Goal Attainment Scale. The goals will concern several aspects of daily life (e.g. to dress up, to brush your teeth). The initial Goal is set at -2 point scale. on Each goal is rated on a 5-point scale: Much less than expected (-2); Somewhat less than expected (-1) ; Expected level of achievement (0); Much more than expected outcome (+2), Somewhat more than expected (+1). A higher score (closer to +2) indicates a better outcome, meaning the goal was achieved beyond expectations. Assessment of the achievement of these goals six months after surgery
Change of hypoxemia before and after surgery | Between 1 month before surgery and 3 months after surgery
  Assessment through night-time oximetry of the number of hypoxemia episodes with oxygen saturation (SpO2 < 90%) and measurement of percentage of time spent in hypoxemia.
  Comparison of the hypoxemia between one month before surgery and six months after surgery.
Change of hypoxemia before and after surgery | Between 1 month before surgery and 6 months after surgery
  Assessment through night-time oximetry of the number of hypoxemia episodes with oxygen saturation (SpO2 < 90%) and measurement of percentage of time spent in hypoxemia.
  Comparison of the hypoxemia between one month before surgery and six months after surgery.
Change of hypercapnia before and after surgery | Between 1 month before surgery and 3 months after surgery
  Assessment through night capnography of the number of hypercapnia episodes (PaCO2 > 50 mmHg) and measurement of percentage of time spent in hypercapnia.
  Comparison of the hypercapnia between one month before surgery and six months after surgery.
Change of hypercapnia before and after surgery | Between 1 month before surgery and 6 months after surgery
  Assessment through night capnography of the number of hypercapnia episodes (PaCO2 > 50 mmHg) and measurement of percentage of time spent in hypercapnia.
  Comparison of the hypercapnia between one month before surgery and six months after surgery.
Change of tidal volume before and after surgery | Between 1 month before surgery and 3 months after surgery
  Assessment of the tidal volume (mL) through spirometry Comparison of the tidal volume between one month before surgery and three months after surgery
Change of tidal volume before and after surgery | Between 1 month before surgery and 6 months after surgery
  Assessment of the tidal volume (mL) through spirometry Comparison of the tidal volume between one month before surgery and three months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No